CLINICAL TRIAL: NCT07237659
Title: A Phase 1a/b, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety of NTR-1011 in Healthy Adults and Adult Patients With Systemic Lupus Erythematosus (SLE) and Rheumatoid Arthritis (RA)
Brief Title: Phase 1a/b Tolerability of NTR-1011 in Healthy Adults and Adult Patients With SLE and RA
Acronym: LIBERATEI
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Neutrolis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NTR1011-001
Record Dates: First submitted 2025-11-12; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: SLE (Systemic Lupus); RA - Rheumatoid Arthritis
Keywords: LIBERATE I; Neutrolis; DNase1L3 fusion protein; DNase1L3 analogue
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Low dose SC NHV (Experimental): Lowest subcutaneous dosage in normal healthy volunteers
  Interventions: Drug: NTR1011
- Mid dose SC NHV (Experimental): middle subcutaneous dosage in normal healthy volunteers
  Interventions: Drug: NTR1011
- High dose SC NHV (Experimental): Highest subcutaneous dosage SC in normal healthy volunteers
  Interventions: Drug: NTR1011
- Low dose IV NHV (Experimental): lowest intravenous dosage in normal healthy volunteers
  Interventions: Drug: NTR1011
- Mid dose IV NHV (Experimental): middle intravenous dosage in normal healthy volunteers
  Interventions: Drug: NTR1011
- High dose IV NHV (Experimental): highest intravenous dosage in normal healthy volunteers
  Interventions: Drug: NTR1011
- Placebo, IV (Placebo Comparator): 0 mg/kg, IV NHV
  Interventions: Drug: NTR1011
- Placebo, SC (Placebo Comparator): 0 mg/kg, SC NHV
  Interventions: Drug: NTR1011

INTERVENTIONS:
Drug: NTR1011 — NTR-1011 will be presented as a solution for subcutaneous (SC) and intravenous (IV) administration.

SUMMARY:
This phase 1a and 1b study is designed to evaluate the safety, tolerability, pharmacokinetics, pharmacodynamics, immunogenicity, and preliminary efficacy of NTR-1011 in healthy adults and in adult patients with systemic lupus erythematosus and rheumatoid arthritis. The main goals of this study are to determine the safety profile of NTR-1011 across subcutaneous and intravenous dose levels, understand how the drug behaves in the body, characterize its biological activity through relevant pharmacodynamic markers, assess the potential for immune responses to treatment, and explore early signals of clinical benefit in autoimmune disease settings.

This is a randomized, double blind, placebo controlled study that begins with a single ascending dose evaluation in healthy volunteers followed by a multiple dose assessment in patients. The design is intended to define the highest safe and well tolerated dose, establish a robust PK and PD baseline, and generate initial patient level evidence to support dose selection and advancement into subsequent clinical development.

ELIGIBILITY:
1. Healthy males and females between 18 and 55 years of age.
2. Body mass index between 17.0 and 30.0 kg/m2.
3. Healthy with no clinically significant findings, as determined by medical evaluation (medical history, physical examination, vital signs, 12-lead electrocardiogram (ECG), and clinical laboratory evaluations) at Screening Visit.
4. Participant voluntarily agrees to participate in this study and signs an Ethics Committee (EC) approved informed consent form (ICF) prior to performing any of the Screening Visit procedures.
5. Participant can understand and is willing to comply with all study requirements, and willing to follow the instructions of the study staff.

Exclusion Criteria:

1. Pregnancy, nursing, and/or breastfeeding.
2. The participant has used an investigational drug within 30 days (or 5 half-lives whichever is longer) before the first dose of the study intervention.

2. Has received any prescription or nonprescription over the counter (except occasional use of acetaminophen, paracetamol, or ibuprofen prior to dosing) medication during the last 14 days. Occasional use is defined at the Investigator's discretion.

3. Has a positive urine test for drugs of abuse, or cotinine at the Screening Visit, regular consumption of alcohol within 6 months before screening or use of illicit substances within 3 months before the Screening Visit.

4. Has a positive test for hepatitis B surface antigen, hepatitis C virus and/or human immunodeficiency virus (HIV).

5. Donation or loss of blood or plasma within 4 weeks before initial dosing.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-09-04 (Actual); Primary Completion 2026-01-07 (Estimated); Study Completion 2026-01-07 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability | 30 days
  Incidence of safety and tolerability (DLTs) to inform RP2D

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Reiff, PhD, MD, Study Chair — Neutrolis; Hakop Gevorkyan, MD, Principal Investigator — California Clinical Trials Medical Group
Locations (1):
- California Clinical Trials Medical Group, Glendale, California, United States

IPD SHARING:
Plan to Share IPD: No
No value outside of this trial